CLINICAL TRIAL: NCT00332969
Title: Efficacy of Medical Treatment With Octreotide in Patients With Primary Inoperable Thymoma to Reduce Tumor Size
Brief Title: Efficacy of Octreotide Treatment in Patients With Primary Inoperable Thymoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSMS995ADE13
Record Dates: First submitted 2006-06-01; First posted 2006-06-02 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2011-11

CONDITIONS: Thymoma
Keywords: Open label; phase II; disease; clinical trial; Octreotide; thymoma; cancer; tumor
MeSH Terms: conditions — Thymoma; Disease; Neoplasms | interventions — Octreotide

ARMS (1):
- Sandostatin (Experimental)
  Interventions: Drug: Octreotide

INTERVENTIONS:
Drug: Octreotide

SUMMARY:
This study will investigate the efficacy of treatment with octroetide in patients with primary inoperable thymoma to reduce tumor size.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged >18 years
2. Inoperability of thymic tumor. Inoperability is defined as at least adherence of the tumor to the neighbour organs, suspicious to infiltrate neighbour organs so that R0 resection cannot be expected.
3. Positive result in SMS-szintigraphy,
4. Thymomas of all WHO based histological subtypes (Rosai, 1999; Travis 2004) at Masaoka stage III based on histological examination of core biopsies or resection specimens.
5. Patients with and without thymoma associated paraneoplastic syndrome
6. Demonstrated tolerance to a test dose of s.c. octreotide injection at Visit 1.

Exclusion Criteria:

1. Performance status 0,1, or 2 (ECOG)
2. Symptomatic cholelithiasis,
3. Pretreatment with octreotide (longn acting release) within the 3 months
4. Patient has received any other investigational agents within 28 days of first day of study drug dosing
5. Patient is < 5 years free of another primary malignancy except: if the other primary malignancy is not currently clinically significant nor requiring active intervention, or if other primary malignancy is a basal cell skin cancer or a cervical carcinoma in situ. Existence of any other malignant disease is not allowed
6. Grade III/IV cardiac problems as defined by the New York Heart Association Criteria. (i.e., congestive heart failure, myocardial infarction within 6 months of study)

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-09; Primary Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Shrinkage of tumor size and diameter of 3 respectively 6 months | 6 months

SECONDARY OUTCOMES:
Resection status after 3 respectively 6 months | 3 - 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (1):
- Novartis Investigative Site, Regensburg, Germany

REFERENCES:
- [Result] Kirzinger L, Boy S, Marienhagen J, Schuierer G, Neu R, Ried M, Hofmann HS, Wiebe K, Strobel P, May C, Kleylein-Sohn J, Baierlein C, Bogdahn U, Marx A, Schalke B. Octreotide LAR and Prednisone as Neoadjuvant Treatment in Patients with Primary or Locally Recurrent Unresectable Thymic Tumors: A Phase II Study. PLoS One. 2016 Dec 16;11(12):e0168215. doi: 10.1371/journal.pone.0168215. eCollection 2016. PMID 27992479